CLINICAL TRIAL: NCT02137746
Title: Open-label, One-arm, Multi-centre Phase II Clinical Trial Treated With Second Cycle of Active Cellular Immunotherapy With DCVAC/PCa in Patients With Localized Prostate Cancer After Primary Radical Prostatectomy Without Objective Progression
Brief Title: Study to Allow for Second Treatment Cycle of DCVAC in Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP010; 2013-003809-26 (EudraCT Number)
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2015-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DCVAC/PCa Arm (Experimental): Dendritic Cells DCVAC/PCa Experimental therapy
  Interventions: Biological: Dendritic Cells DCVAC/PCa

INTERVENTIONS:
Biological: Dendritic Cells DCVAC/PCa — DCVAC/PCa Experimental therapy

SUMMARY:
The purpose of this study is to assess the safety of the second cycle of DCVAC/PCa in patients who completed the first cycle of DCVAC/PCa in the clinical trial SP003 without an objective progression of the disease.

DETAILED DESCRIPTION:
Same as brief summary

ELIGIBILITY:
Inclusion Criteria:

* Male 18 years and older
* Histologically confirmed prostate adenocarcinoma Stage pathological tumor-2 (pT2)
* Post radical Primary Prostatectomy
* Completion of DCVAC/PCa arm in Study SP003, without objective progression of the disease

Exclusion Criteria:

* Prior androgen deprivation therapy for prostate cancer
* Peripheral neuropathy of Common Toxicity Criteria (CTC) grade 2 or greater
* Other uncontrolled intercurrent illness
* Treatment with immunotherapy against PCa
* Clinically significant cardiovascular disease
* Active autoimmune disease requiring treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Safety evaluation of the second cycle of DCVAC | 52 weeks
  Safety evaluation of the second cycle of active cellular immunotherapy, which includes a second leukapheresis procedure, who after primary radical prostatectomy completed first cycle of active cellular immunotherapy in clinical trial SP003 without objective disease progression requiring additional anti-tumor therapy.

SECONDARY OUTCOMES:
Time to Prostate Specific Antigen (PSA) Doubling Time | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Scheiner, PhD, Study Director — Sotio Biotech Inc.
Locations (7):
- Czechia (7):
  - Hradec Králové
  - Jablonec nad Nisou
  - Nový Jičín
  - Olomouc
  - Prague
  - Uherské Hradiště
  - Ústí nad Labem